CLINICAL TRIAL: NCT02485275
Title: Stroke Imaging Package Study
Acronym: SIPS
Status: Completed | Type: Observational
Sponsor: Wei-Hai Xu (Other)
Collaborators: Peking Union Medical College Hospital (Other); The Third Medical Center of Chinese PLA General Hospital (Unknown); Army Medical Center of PLA (Other Government); The General Hospital of Northern Theater Command (Other); Subei People's Hospital of Jiangsu Province (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Beijing Jishuitan Hospital (Other); Fujian Medical University Union Hospital (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of University of South China (Other); Qilu Hospital of Shandong University (Other); Tangshan Gongren Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Renmin Hospital of Wuhan University (Other); China-Japan Union Hospital, Jilin University (Other); Shanghai Tong Ren Hospital (Other)
Responsible Party: Sponsor-Investigator, Wei-Hai Xu, Associate Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: HRMRI
Record Dates: First submitted 2015-06-25; First posted 2015-06-30 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Acute Ischemic Stroke; Intracranial Arteriosclerosis; Cerebral Small Vessel Diseases
Keywords: AIS; ICAS; CSVD
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis; Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Our study aims to explore the value of new imaging technique package in predicting early neurological deterioration (END) as well as 90-day unfavorable outcome in patients with acute ischaemic stroke.

DETAILED DESCRIPTION:
1. Patients with acute ischemic stroke within 4.5-72h after onset were prospectively enrolled in our study and underwent standardized clinical and new imaging technique package assessment.
2. New imaging technique package mainly includes conventional cranial MRI （T1,T2,T2 FLAIR,DWI, and ADC), cranial magnetic resonance angiography (MRA), and intracranial vessel wall imaging (High-Resolution Magnetic Resonance Imaging,HRMRI) as well as susceptibility weighted imaging (SWI).
3. The neurofunctional fluctuation during hospitalization as well as 90-day outcomes were carefully assessed. Patients were followed up for 90-days after stroke onset.
4. Our study aims to explore the value of new imaging technique package in predicting early neurological deterioration (END) as well as 90-day unfavorable outcome in patients with acute ischaemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. patients with ischemic stroke and hospitalized during 4.5-72 hours after onset , confirmed by diffusion weighted imaging (DWI).
2. patients with stable vital signs.
3. patients who have underwent thrombolytic/intravascular therapy are allowed to enroll in the study.

Exclusion Criteria:

1. patients with absolute/relative contraindication to MRI (including but not confined to metal in the body and claustrophobia).
2. patients who is extremely agitated, and cannot comply with MRI exam.
3. patients who declined the consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the collaborative stroke centers and will be followed for the duration of their hospitalization. Patients will be followed up until at least 3 months after stroke onset.
Sampling Method: Non-Probability Sample
Enrollment: 949 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
early neurological deterioration within 3 weeks after stroke onset (END-3 weeks) | 3 weeks after stroke onset
  END-3 weeks is defined as a significant neuro-functional decline [increment of the National Institutes of Health Stroke Scale (NIHSS) ≥ 2 points ] within 3 weeks after admission.
90-days prognosis | 90-days after stroke onset
  90-days prognosis included two parts :1) stroke recurrence with new lesion on DWI;2) the modified Ranking Score (mRS) at 90-days after stroke onset.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - The Third Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Army Medical Center of PLA, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Qingdao, Shandong
  - Tongren Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Background] Mazighi M, Labreuche J, Gongora-Rivera F, Duyckaerts C, Hauw JJ, Amarenco P. Autopsy prevalence of intracranial atherosclerosis in patients with fatal stroke. Stroke. 2008 Apr;39(4):1142-7. doi: 10.1161/STROKEAHA.107.496513. Epub 2008 Feb 28. PMID 18309170
- [Background] Li ML, Xu WH, Song L, Feng F, You H, Ni J, Gao S, Cui LY, Jin ZY. Atherosclerosis of middle cerebral artery: evaluation with high-resolution MR imaging at 3T. Atherosclerosis. 2009 Jun;204(2):447-52. doi: 10.1016/j.atherosclerosis.2008.10.019. Epub 2008 Oct 25. PMID 19041971
- [Background] Xu WH, Li ML, Gao S, Ni J, Zhou LX, Yao M, Peng B, Feng F, Jin ZY, Cui LY. In vivo high-resolution MR imaging of symptomatic and asymptomatic middle cerebral artery atherosclerotic stenosis. Atherosclerosis. 2010 Oct;212(2):507-11. doi: 10.1016/j.atherosclerosis.2010.06.035. Epub 2010 Jun 25. PMID 20638663
- [Background] Xu WH, Li ML, Gao S, Ni J, Zhou LX, Yao M, Peng B, Feng F, Jin ZY, Cui LY. Plaque distribution of stenotic middle cerebral artery and its clinical relevance. Stroke. 2011 Oct;42(10):2957-9. doi: 10.1161/STROKEAHA.111.618132. Epub 2011 Jul 28. PMID 21799160
- [Background] Xu WH, Li ML, Gao S, Ni J, Yao M, Zhou LX, Peng B, Feng F, Jin ZY, Cui LY. Middle cerebral artery intraplaque hemorrhage: prevalence and clinical relevance. Ann Neurol. 2012 Feb;71(2):195-8. doi: 10.1002/ana.22626. PMID 22367991
- [Background] Xu WH, Li ML, Niu JW, Feng F, Jin ZY, Gao S. Intracranial artery atherosclerosis and lumen dilation in cerebral small-vessel diseases: a high-resolution MRI Study. CNS Neurosci Ther. 2014 Apr;20(4):364-7. doi: 10.1111/cns.12224. Epub 2014 Jan 15. PMID 24423003
- [Background] Xu WH, Li ML, Niu JW, Feng F, Jin ZY, Gao S. Deep tiny flow voids along middle cerebral artery atherosclerotic occlusions: a high-resolution MR imaging study. J Neurol Sci. 2014 Apr 15;339(1-2):130-3. doi: 10.1016/j.jns.2014.01.042. Epub 2014 Feb 6. PMID 24530171
- [Background] Li M, Wu SW, Xu WH. High-resolution MRI of radiation-induced intracranial vasculopathy. Neurology. 2015 Feb 10;84(6):631. doi: 10.1212/WNL.0000000000001223. No abstract available. PMID 25666631
- [Derived] Zhang ZM, Si QQ, Chen HS, Yang Y, Zhang M, Wu SW, Meng Y, Li ML, Lin QQ, Liebeskind DS, Huang YN, Xu WH. High-resolution magnetic resonance imaging of acute intracranial artery thrombus. Eur J Neurol. 2023 Oct;30(10):3172-3181. doi: 10.1111/ene.15985. Epub 2023 Aug 7. PMID 37452734